CLINICAL TRIAL: NCT04105933
Title: The Effects of Culturally Sensitive Cognitive Behavioural Therapy on Women Experienced Intimate Partner Violence
Brief Title: Culturally Sensitive Cognitive Behavioural Therapy for the Survivors of Intimate Partner Violence (IPV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/013298
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-09

CONDITIONS: Mental Abuse of Adult; Emotional Abuse; Domestic Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS-CBT (Experimental): Culturally sensitive-CBT intervention was comprised of 16 sessions of cognitive behavioral therapy focused on culturally-specific beliefs and attitude.
  Interventions: Other: CS-CBT
- CBT (Active Comparator): CBT intervention was comprised of 16 sessions of cognitive behavioral therapy.
  Interventions: Other: CBT

INTERVENTIONS:
Other: CS-CBT — Culturally sensitive Cognitive Behavioural Therapy was delivered individually, focused on potential cultural beliefs and attitudes that might collide with core values of CBT.
  Arms: CS-CBT
Other: CBT — CBT was delivered at an individual level, dealing with thoughts, feelings and behaviours in the present. Thoughts are identified and then challenged, to make them more objective and rational.
  Arms: CBT

SUMMARY:
Women experience negative psychological outcomes long after the violent relationship has ended. Women suffer constant trauma and psychological distress being in emotional and mentally abusive relationship. Present study developed Culturally sensitive cognitive-behaviour therapy (CBT) to fit the client's cultural identity, context, and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Women victim of intimate partner violence
* Still in relationship with abuser
* Willing to attend 16-weeks sessions

Exclusion Criteria:

* In need of clinical supervision or treatment
* Severe mental disorders
* Cognitive disorders
* Refused to give written consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-02-11 (Actual)

PRIMARY OUTCOMES:
Psychological symptoms | Change from baseline to 16 weeks
  Brief Symptom Inventory (BSI) was used to assess psychological complaints

SECONDARY OUTCOMES:
Self esteem | Change from baseline to 16 weeks
  Rosenberg Self-Esteem Scale was used to assess self esteem
Forgiveness | Change from baseline to 16 weeks
  Heartland Forgiveness Scale was used to assess forgiveness to oneself, to other and to situation

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Warwick Research Services; Rachana Khandelwal, PhD, Study Chair — NMP Medical Research Institute, India; Anurag Sharma, MPhil, Principal Investigator — Patan Girls College, India
Locations (2):
- India (2):
  - Gyansaneejvani, Būndi, Rajasthan
  - NMP Medical Research Institute, Jaipur, Rajasthan